CLINICAL TRIAL: NCT05639868
Title: Is Video-assisted Cardiopulmonary Resuscitation More Effective Than Telephone-assisted or Not-instructed Cardiopulmonary Resuscitation by Laypeople? - a Randomized Controlled Simulation Study
Brief Title: Effectiveness of Video-assisted Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr. Bálint Bánfai, senior lecturer, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Upecs_V-CPR
Record Dates: First submitted 2022-11-14; First posted 2022-12-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-CPR (Active Comparator): Participants perform telephone-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Other: Video-assisted CPR; Other: Telephone-assisted CPR
- V-CPR (Experimental): Participants perform video-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Other: Video-assisted CPR; Other: Telephone-assisted CPR
- Unassisted CPR (No Intervention): CPR without dispatcher instructions.

INTERVENTIONS:
Other: Video-assisted CPR — Participants in V-CPR group get video-based (vocal and visual) instructions from the dispatcher.
  Arms: T-CPR; V-CPR
Other: Telephone-assisted CPR — Participants in T-CPR group get voice-based (vocal) instructions from the dispatcher.
  Arms: T-CPR; V-CPR

SUMMARY:
Sudden cardiac arrest is a major public health problem worldwide and it is one of the leading causes of death in industrialized countries. Emergency Medical Services (EMS) dispatchers play an important role to recognize cardiac arrest and give help to the lay first responder via telephone CPR (T-CPR) which improves survival rates. The current technology allows the live video connection between the scene and the dispatcher which provides the opportunity for video-assisted CPR (V-CPR) via the bystander smartphone.

Effectiveness of V-CPR has only been investigated to a limited extent. Comparing effectiveness of V-CPR (effectiveness of chest compression, time parameters eg. time to first chest compression) to T-CPR and non-instructed CPR can be useful to implement V-CPR technology.

DETAILED DESCRIPTION:
Sudden cardiac arrest is a major public health problem worldwide and it is one of the leading causes of death in industrialized countries. EMS dispatchers play an important role to recognize cardiac arrest and give help to the lay first responder via telephone CPR (T-CPR) which improves survival rates. The current technology allows the live video connection between the scene and the dispatcher which provides the opportunity for video-assisted CPR (V-CPR) via the bystander smartphone.

Effectiveness of V-CPR has only been investigated to a limited extent. Comparing effectiveness of V-CPR (quality of chest compressions: depth, rate, hand position), time parameters: time to recognize cardiac arrest, time of check breathing, total no-flow time, to first chest compression) to T-CPR and non-instructed CPR can be useful to implement V-CPR technology.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* healthcare professionals (paramedics, nurses, etc.)
* pregnant women
* people with cardio-pulmonary and musculoskeletal diseases or any other impairment that would risk harm for the volunteer while performing CPR for 2 minutes
* psychological disabilities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Quality of chest compressions (depth of chest compressions). | During procedure
  Chest compression depth will be evaluated by a manikin connected to a CPR software.
Quality of chest compressions (rate of chest compressions). | During procedure
  Chest compression rate will be evaluated by a manikin connected to a CPR software.
Quality of chest compressions (hand position of chest compressions). | During procedure
  Hand position during chest compression will be evaluated by observation.

SECONDARY OUTCOMES:
Time factors of CPR | During procedure
  Measuring the time of check breathing, time to recognize cardiac arrest, time to first chest compression, and cumulative time of no-flow time by the CPR software and observation.
Attitude of bystanders. | Immediately after the CPR procedure (within 15 minutes)
  Subjective feelings after performing CPR based on a short survey using Likert-scale based queries (lower numbers indicate worse, higher score indicates better opinion).

CONTACTS AND LOCATIONS:
Overall Officials: Bálint Bánfai, PhD, Principal Investigator — University of Pecs
Locations (1):
- University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szollosi V, Horvath B, Nemeth D, Banfai-Csonka H, Betlehem J, Banfai B. A randomized controlled simulation trial comparing video-assisted with telephone-assisted and unassisted cardiopulmonary resuscitation performed by non-healthcare university students. Sci Rep. 2023 Sep 11;13(1):14925. doi: 10.1038/s41598-023-42131-z. PMID 37696968